CLINICAL TRIAL: NCT02105987
Title: 201147: a Phase IIIb, Randomized, Open-label Study of the Safety, Efficacy, and Tolerability of Switching to a Fixed-dose Combination of Abacavir/Dolutegravir/ Lamivudine From Current Antiretroviral Regimen Compared With Continuation of the Current Antiretroviral Regimen in HIV-1 Infected Adults Who Are Virologically Suppressed, The STRIIVING Study.
Brief Title: A Phase IIIb Study of the Safety, Efficacy, and Tolerability of Switching to a Fixed-dose Combination of Abacavir/Dolutegravir/ Lamivudine From Current Antiretroviral Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: PPD Development, LP (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201147; NCT02131025 (obsolete NCT alias)
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Abacavir/dolutegravir/lamivudine; Fixed-dose combination; Once daily; Trii; Single-tablet regimen
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABC/DTG/3TC (Experimental): Subject will take ABC 600 mg/DTG 50 mg/3TC 300 mg FDC once daily in the morning or the evening, at approximately the same time each day for 24 weeks. After Week 24, subjects will continue on this treatment arm for an additional 24 weeks.
  Interventions: Drug: ABC/DTG/3TC FDC
- Comparator (Active Comparator): Subjects will continue on their current Combination antiretroviral therapy (cART) regimen for 24 weeks. At Week 24, subjects will switch to ABC/DTG/3TC FDC for an additional 24 weeks.
  Interventions: Drug: Ongoing cART regimen

INTERVENTIONS:
Drug: ABC/DTG/3TC FDC — Purple, oval, biconvex tablets containing 702 mg Abacavir sulphate which is equivalent to 600 mg ABC, 52.62 mg Dolutegravir sodium which is equivalent to 50 mg Dolutegravir free acid and 300 mg 3TC
  Arms: ABC/DTG/3TC
Drug: Ongoing cART regimen — Stable cART regimens including boosted PI (or ATV unboosted) + 2 NRTIs; NNRTI + 2 NRTIs, or INI (RAL or EVG)+ 2 NRTIs
  Arms: Comparator

SUMMARY:
This study is a 48-week, Phase IIIb, randomly assigned, open-label, active-controlled, multicenter, parallel group, non-inferiority study. This study is designed to demonstrate the non-inferior antiviral activity of switching to the Abacavir (ABC) 600 milligrams (mg)/Dolutegravir(DTG) 50 mg/Lamivudine (3TC) 300 mg fixed-dose combination (FDC) compared with continuing the subject's current suppressive regimen through 24 weeks. The study will be conducted in approximately 538 Human Immunodeficiency Virus -1 (HIV-1) infected individuals who are on stable suppressive combination antiretroviral therapy (cART) with 2 Nucleoside reverse transcriptase inhibitors (NRTIs) plus either a protease inhibitor (PI), an non-nucleoside reverse transcriptase inhibitor (NNRTI), or an integrase inhibitor (INI). Eligible subjects will be randomly assigned 1:1 to continue their current regimen (approximately 269 subjects) or be switched to ABC/DTG/3TC FDC (approximately 269 subjects) once daily for 24 weeks. At Week 24, individuals originally randomly assigned to continue their current regimen will switch to ABC/DTG/3TC FDC and be followed for an additional 24 weeks. Individuals initially randomly assigned to ABC/DTG/3TC FDC will continue on that treatment arm for an additional 24 weeks. A pharmacokinetic (PK) substudy will be conducted at a small number of sites (approximately 10) to evaluate predose DTG concentrations as well as residual drug concentrations of efavirenz (EFV), nevaripine (NVP), amprenavir (APV) and tipranavir (TPV) in a subgroup of subjects who switch from EFV, NVP, fosamprenavir/ritonavir (FPV/r) or tipranavir/ritonavir (TPV/r).

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand and comply with protocol requirements, instructions, and restrictions;
* Be likely to complete the study as planned;
* Be considered appropriate candidates for participation in an investigative clinical trial with oral medication (e.g., no active substance abuse, acute major organ disease, or planned long-term work assignments out of the country, etc.).
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening
* HIV-1 infected men or women >=18 years of age;
* A female may be eligible to enter and participate in the study if she: a. Is of non-childbearing potential either defined as post-menopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy, or bilateral oophorectomy or,
* A female may be eligible to enter and participate in the study if she: b. Is of childbearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy: Complete abstinence from intercourse from 2 weeks prior to administration of study drug, throughout the study, and for at least 2 weeks after discontinuation of all study drugs; Double barrier method (e.g., male condom/spermicide, male condom/diaphragm, diaphragm/spermicide); Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year ; Male partner sterilization prior to the female subject's entry into the study and this male is the sole partner for that subject; Approved hormonal contraception for subjects randomly assigned to the ABC/DTG/3TC arm or approved hormonal contraception plus a barrier method for subjects assigned to continued antiretroviral therapy arm; Any other method with published data showing that the expected failure rate is <1% per year.
* Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of study drug. A childbearing potential female subject who starts the study using complete abstinence as her contraceptive method and decides to become sexually active must use the double barrier method either as a bridge to an approved hormonal contraception (if possible) or as a method of choice to be maintained from that moment onwards.
* All subjects participating in the study should be counselled on safer sexual practices including the use of effective barrier methods (e.g., male condom/spermicide).
* Within the last year, 2 consecutive plasma HIV-1 Ribonucleic acid (RNA) measurements <50 copies/millilitres (c/mL) and plasma HIV-1 RNA<50 c/mL at Screening (<75 b Deoxyribonucleic acid [bDNA] is considered equal to <50 c/mL); Subjects who present at initial screening with a viral load between 50 to 200 c/mL can be retested once within the screening period.
* Must be on current regimen (whether first or second line Combination antiretroviral therapy [cART]) for at least 6 months prior to Screening;
* Acceptable stable cART regimens prior to Screening include: • Boosted PI (or Atazanavir [ATV]) unboosted) + 2 NRTIs, NNRTI + 2 NRTIs, • INI + 2 NRTIs. For subjects on an INI, their INI at Screening must be RAL or Elvitegravir (EVG)
* Any switch to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability and/or safety concerns.
* Subject must have achieved plasma HIV-1 RNA level <50 c/mL within 6 months of start of initial cART regimen with no plasma HIV-1 RNA level >200 c/mL following initial suppression;
* Documentation that the subject is negative for the human leukocyte antigen (HLA) B*5701 allele;

Exclusion Criteria:

Exclusionary Medical Conditions

* Women who are breastfeeding;
* Any evidence of an active (Centers for Disease Control and Prevention [CDC] Category C) disease. Exceptions include cutaneous Kaposi's sarcoma not requiring systemic therapy and historic CD4+ cell counts of <200 cells/cubic millimeter (mm).
* Subjects with any degree of hepatic impairment;
* Subjects positive for hepatitis B virus surface antigen (+HBsAg) at Screening or with an anticipated need for hepatitis C virus (HCV) therapy during the study;
* History or presence of allergy to the study drugs or their components or drugs of their class;
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the study medical monitor for inclusion of the subject;
* Subjects who, in the investigator's judgment, pose a significant suicidality risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk;

Exclusionary Treatments Prior to Screening or Day 1

* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening;
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any immunomodulators that alter immune responses;
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study drug;
* A history of use of only mono or dual NRTI therapy prior to starting cART;
* Use of etravirine at time of switch;
* Use of DTG at time of switch;
* Subjects receiving any prohibited medication listed in the protocol and who are unwilling or unable to switch to an alternate medication

Exclusionary Laboratory Values or Clinical Assessments at Screening

* Evidence of primary viral resistance based on the presence of any resistance-associated major PI or any NRTI, NNRTI, or INI mutation in any prior resistance genotype assay result;
* Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 triglyceride abnormalities. A single repeat test is allowed during the screening period to verify a result;
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the subject's participation in the study of an investigational compound;
* Alanine aminotransferase (ALT) >=5 times the upper limit of normal (ULN), or ALT >=3 × ULN and bilirubin >=1.5 × ULN (with >35% direct bilirubin);
* Subject has CrCl of <50 mL/min using Modification of Diet in Renal Disease (MDRD);
* QTc (Bazett) >=450 msec or QTc (Bazett) >=480 msec for subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB). The QTc should be based on a single QTc value electrocardiogram (ECG) obtained.
* Eligibility of subjects for study participation will be decided by the investigators after taking into consideration various country specific guidelines, and notwithstanding the above mentioned minimum inclusion and exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (77):
- United States (67):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Seattle, Washington
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Puerto Rico (4):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, Rio Piedras, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
  - GSK Investigational Site, San Juan

REFERENCES:
- [Derived] Trottier B, Lake JE, Logue K, Brinson C, Santiago L, Brennan C, Koteff JA, Wynne B, Hopking J, Granier C, Aboud M. Dolutegravir/abacavir/lamivudine versus current ART in virally suppressed patients (STRIIVING): a 48-week, randomized, non-inferiority, open-label, Phase IIIb study. Antivir Ther. 2017;22(4):295-305. doi: 10.3851/IMP3166. Epub 2017 Apr 12. PMID 28401876

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 841 participants (par.) were screened and 555 human immunodeficiency virus type 1 (HIV-1) infected par. who were on stable suppressive combination antiretroviral therapy (cART) with 2 nucleoside reverse transcriptase inhibitor (NRTIs) plus either a protease inhibitor (PI), an non-NRTI (NNRTI), or an integrase inhibitor (INI) were randomized.
Groups:
- ABC 600 mg / DTG 50 mg /3TC 300 mg FDC: Participants received abacavir (ABC) 600 milligrams (mg)/ dolutegravir (DTG) 50 mg/ lamivudine (3TC) 300 mg fixed-dose combination (FDC) tablets with or without food once daily in the morning or the evening at approximately the same time each day for 24 weeks.
- Current ART: Participants continued on their current ART regimen for 24 weeks.
- ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch: Participants who completed early switch phase continued to receive ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablets with or without food once daily in the morning or the evening at approximately the same time each day for an additional 24 weeks.
- ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch: Participants who completed early switch phase and maintained viral suppression (<50 Copies per milliliter [c/mL]) were switched to ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablets and were followed for an additional 24 weeks of treatment.
- ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch:Cont Phase; ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch:Cont Phase: If ABC/DTG/3TC was not locally approved and commercially available when a participant successfully completed the Week 48 visit, the participant had the opportunity to enter into the Continuation Phase. During the Continuation Phase, participants were supplied with ABC/DTG/3TC until it was locally approved and commercially available.
Period: Early Switch Phase (24 Weeks)
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch:Cont Phase | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch:Cont Phase
Started | 275 (Number Started represents the number of par. in the Intent-To-Treat Exposed (ITT-E) Population.) | 278 (Number Started represents the number of par. in the Intent-To-Treat Exposed (ITT-E) Population.) | 0 | 0 | 0 | 0
Completed | 239 | 244 | 0 | 0 | 0 | 0
Not Completed | 36 | 34 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 15 | 17 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Missing Disposition Data | 0 | 1 | 0 | 0 | 0 | 0
Period: Late Switch Phase (24 Weeks)
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch:Cont Phase | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch:Cont Phase
Started | 0 | 0 | 275 | 244 | 0 | 0
Completed | 0 | 0 | 230 | 230 | 0 | 0
Not Completed | 0 | 0 | 45 | 14 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 10 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 15 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 8 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 5 | 0 | 0 | 0
Not completed — met protocol defined stopping criteria | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Per sponsor request | 0 | 0 | 1 | 0 | 0 | 0
Period: Continuation Phase
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Early Switch:Cont Phase | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC Late Switch:Cont Phase
Started | 0 | 0 | 0 | 0 | 14 | 23
Completed | 0 | 0 | 0 | 0 | 13 | 23
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Early Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC: Participants received ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablets with or without food once daily in the morning or the evening at approximately the same time each day for 24 weeks. At Week 24, participants will continue on this treatment for an additional 24 weeks.
- Late Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC: Participants continued on their current ART regimen for 24 weeks. At Week 24, participants originally randomly assigned to continue their current regimen switched to ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablets and were followed for an additional 24 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | Early Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Late Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Total
Number analyzed (Participants) | 275 | 244 | 519
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (10.61) | 45.5 (11.25) | 44.8 (10.93)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 32 | 70
  Male | 237 | 212 | 449
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 81 | 63 | 144
  American Indian or Alaska Native | 3 | 2 | 5
  Asian - Central/South Asian Heritage | 1 | 2 | 3
  Asian - East Asian Heritage | 1 | 3 | 4
  Asian - Japanese Heritage | 1 | 1 | 2
  Asian - South East Asian Heritage | 1 | 2 | 3
  Asian - Mixed Race | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 1 | 2
  White - Arabic/North African Heritage | 2 | 0 | 2
  White - White/Caucasian/European Heritage | 176 | 165 | 341
  White - Mixed Race | 3 | 3 | 6
  White - Asian | 1 | 1 | 2
  Mixed Race | 1 | 1 | 2
  Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) <50 Copies Per Milliliter (c/mL) at Week 24 Using the Snapshot Algorithm
Description: The Food and Drug Administration (FDA) snapshot (Missing, Switch or Discontinuation = Failure) algorithm is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy. Virologic Success (e.g., <50 c/mL) or virologic failure within an analysis window is typically determined by the last available HIV-1 RNA measurement in that window and in the treatment phase of interest (e.g., Week 24 snapshot outcomes of the early switch phase will not use HIV-1 RNA data from the late switch phase, even if such data is within the Week 24 analysis window). A virologic failure occurs when a participant changes to their ART regimen (e.g., addition of other ARTs to the study-specified regimens, or switches in components of the current ART regimen).
Time Frame: Week 24
Population: Intent-to-Treat Exposed (ITT-E) Population: all participants randomized to ABC/DTG/3TC and receive at least one dose of study drug or randomized to remain on current ART regimen and continue in the study past Day 1.
Measure: Number; unit: Participants
Groups:
- ABC 600 mg / DTG 50 mg /3TC 300 mg FDC: Participants received ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablets with or without food once daily in the morning or the evening at approximately the same time each day for 24 weeks. At Week 24, participants will continue on this treatment for an additional 24 weeks.
- Current ART: Participants continued on their current ART regimen for 24 weeks. At Week 24, participants originally randomly assigned to continue their current regimen switched to ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablets and were followed for an additional 24 weeks of treatment.
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 275 | 278
Participants | 233 | 245
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is -10%; Cochran-Mantel-Haenszel; Mean Difference (Net) = -3.4, 95% CI 2-sided [-9.1 to 2.4] — Based on Cochran-Mantel Haenszel stratified analysis adjusting for the following Baseline stratification factor: Original ART third agent class (PI, NNRTI, or INI)

2. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Counts at Week 24
Description: Change from Baseline in CD4+ cell counts were assessed at Baseline, Weeks 4, 8, 16 and 24. No imputation for missing data or premature discontinuation was performed and the observed values were used. Baseline value is defined as the last pre-treatment value observed. Change from Baseline was calculated as the observed value minus the Baseline value. The Week 24 data were summarized.
Time Frame: Baseline and Week 24
Population: ITT-E Population. Only participants with non-missing CD4 data at Week 24 are included.
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 238 | 248
Cells per cubic millimeter (cells/mm^3) | 50.0 [-48.0 to 130.0] | 11.0 [-60.0 to 103.5]

3. Secondary Outcome: Number of Participants in the Virologic Non-response Category From the Snapshot Analysis at Week 24
Description: Virologic non-responders were defined as the participants with a viral load >=50 c/mL in the Week 24 analysis window. Virologic non-response includes participants who had HIV-1 RNA >=50 c/mL, who discontinued for lack of efficacy, who discontinued for other reasons while not suppressed, data in window but not <50 c/mL, and who changed ART regimen at Week 24. Difference is calculated as the proportion on ABC/DTG/3TC - proportion on current ART regimen.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 275 | 278
Participants | 3 | 4
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.0 to 1.4] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) up to 24 Weeks
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, based on medical or scientific judgment and all events of possible drug-induced liver injury with hyperbilirubinemia. The DAIDS table for grading the severity of adult and pediatric AEs was utilized for AE reporting. The DAIDS estimates the severity grade as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life threatening) for each parameter.
Time Frame: Baseline and up to 24 weeks
Population: Safety Population: all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Participants
  Any AEs | 183 | 129
  Any SAEs | 6 | 5

5. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Chemistry Toxicities up to 24 Weeks
Description: The number of participants with maximum post-Baseline emergent chemistry toxicities for each grade were summarized by parameter. A toxicity is considered emergent if it develops or increases in intensity from Baseline. For participants who were originally randomized to current ART regimen on Day 1 and then switched to ABC/DTG/3TC on Week 24, Baseline is defined as the last non-missing value from the early switch phase and maximum post-Baseline emergent during the late switch phase was determined relative to this Baseline. The DAIDS table for grading the severity of adult and pediatric AEs was utilized for AE reporting. The DAIDS defined the severity grade as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life threatening) for each parameter.
Time Frame: Baseline and up to 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Participants
  Grade 1 | 98 | 108
  Grade 2 | 73 | 71
  Grade 3 | 21 | 25
  Grade 4 | 10 | 10

6. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities up to 24 Weeks
Description: The number of participants with maximum post-Baseline emergent hematology toxicities for each grade were summarized by parameter. A toxicity is considered emergent if it develops or increases in intensity from Baseline. For participants who were originally randomized to current ART regimen on Day 1 and then switched to ABC/DTG/3TC on Week 24, Baseline is defined as the last non-missing value from the early switch phase and maximum post-Baseline emergent during the late switch phase was determined relative to this Baseline. The DAIDS table for grading the severity of adult and pediatric AEs was utilized for AE reporting. The DAIDS defined the severity grade as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life threatening) for each parameter.
Time Frame: Baseline and up to 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Participants
  Grade 1 | 19 | 15
  Grade 2 | 3 | 6
  Grade 3 | 0 | 2
  Grade 4 | 1 | 0

7. Secondary Outcome: Number of Participants With AEs Leading to Withdrawal Over 24 Weeks
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, based on medical or scientific judgment and all events of possible drug-induced liver injury with hyperbilirubinemia.
Time Frame: Baseline and up to 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Participants | 11 | 0

8. Secondary Outcome: Change From Baseline in Fasting Lipids (Cholesterol, LDL Cholesterol, HDL Cholesterol, and Triglycerides) at Week 24
Description: Change from Baseline for each fasting lipid parameters included cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides. Adjusted mean is the estimated mean change from Baseline in each parameter at Week 24 in each arm calculated from an analysis of covariance (ANCOVA) model which includes the following covariates: treatment, original ART third agent class, interaction of treatment and original ART 3rd agent, use of lipid modifying agent and Baseline lipid level. Difference is calculated as ABC/DTG/3TC - Current ART regimen. For fasting lipid assessments, an overnight fast is preferred; however, a minimum of a 6-hour fast was acceptable for participants with afternoon appointments.
Time Frame: Baseline and Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimoles per liter (mmol/L)
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Millimoles per liter (mmol/L)
  Cholesterol,n=226, 231 | 0.10 [0.00 to 0.21] | -0.01 [-0.11 to 0.10]
  LDL Cholesterol, n=221, 226 | 0.10 [0.01 to 0.18] | 0.02 [-0.06 to 0.11]
  HDL Cholesterol, n=226, 231 | 0.00 [-0.04 to 0.03] | -0.03 [-0.06 to 0.01]
  Triglycerides, n=226, 231 | 0.07 [-0.07 to 0.21] | -0.04 [-0.17 to 0.10]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.096, ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.02 to 0.23] — Statistical analysis of cholesterol is presented
Statistical Analysis 2: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.167, ANCOVA; Median Difference (Final Values) = 0.07, 95% CI 2-sided [-0.03 to 0.18] — Statistical analysis of LDL cholesterol is presented
Statistical Analysis 3: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.317, ANCOVA; Median Difference (Final Values) = 0.02, 95% CI 2-sided [-0.02 to 0.06] — Statistical analysis of HDL cholesterol is presented
Statistical Analysis 4: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.187, ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.05 to 0.27] — Statistical analysis of triglycerides is presented

9. Secondary Outcome: Change From Baseline in Fasting Lipids (Total Cholesterol/HDL Cholesterol Ratio) at Week 24
Description: Change from Baseline for fasting lipid parameter total cholesterol/HDL cholesterol ratio. Adjusted mean is the estimated mean change from Baseline at Week 24 in each arm calculated from an analysis of covariance (ANCOVA) model which includes the following covariates: treatment, original ART third agent class, interaction of treatment and original ART 3rd agent, use of lipid modifying agent and Baseline lipid level. Difference is calculated as ABC/DTG/3TC - Current ART regimen. For fasting lipid assessments, an overnight fast is preferred; however, a minimum of a 6-hour fast was acceptable for participants with afternoon appointments.
Time Frame: Baseline and Week 24
Population: Safety Population. Only those participants available at the specified time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 226 | 231
Ratio | 0.10 [-0.02 to 0.22] | 0.00 [-0.12 to 0.12]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.175, ANCOVA; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.04 to 0.25] — Statistical analysis of total cholesterol/HDL cholesterol ratio is presented

10. Secondary Outcome: Change From Baseline in Treatment Satisfaction at Week 4 and Week 24
Description: The HIV treatment satisfaction questionnaire (TSQ) is a 10 item self-reported scale. Individual item scores range from 6 (very satisfied) to 0 (very dissatisfied). The treatment satisfaction total score (range 0-60) is the sum of all the 10 individual items. The general satisfaction/Clinical subscale (range 0-30) is the sum of the 5 clinical items and the lifestyle/ease subscale (range 0-30) is the sum of the remaining 5 lifestyle items. Last observation carried forward (LOCF) were used for the analysis. If a participant had a missing value at Week 24, his previous non-missing available value while on the same treatment was carried forward (ie the Week 4 or withdrawal value is used in the Week 24 summary for participants in the ABC/DTG3TC with missing Week 24 value). Data were analyzed using an ANCOVA model with factors including treatment, Baseline score and stratification factor. Treatment group difference (ABC/DTG/3TC-cART) estimate and 95% CI were presented.
Time Frame: Baseline, Week 4 and Week 24
Population: ITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 275 | 278
Units on a scale
  Total score, n=270,276 | 3.2 (0.40) | 0.8 (0.39)
  General Satisfaction/Clinical Subscale, n=269, 276 | 1.3 (0.24) | 0.2 (0.23)
  Lifestyle/Ease Subscale Score, n=269, 276 | 1.8 (0.19) | 0.6 (0.19)
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 2.4, 95% CI 2-sided [1.3 to 3.5] — Statistical analysis for total score is presented
Statistical Analysis 2: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Net) = 1.0, 95% CI 2-sided [0.4 to 1.7] — Statistical analysis for general satisfaction/clinical subscale score is presented
Statistical Analysis 3: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 1.3, 95% CI 2-sided [0.8 to 1.8] — Statistical analysis for lifestyle/ease subscale is presented

11. Secondary Outcome: Change From Baseline in Creatinine at Week 24
Description: Renal markers included creatinine and summarized based on an observed case (OC) data set at Week 24. Adjusted mean is the estimated mean change from Baseline in each biomarker at Week 24 in each arm calculated from an ANCOVA analysis of covariance model including the following covariates: treatment, original ART third agent class, interaction of treatment and original ART third agent class, and Baseline biomarker level. Differences are calculated as ABC/DTG/3TC - Current ART regimen.
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Micromoles per liter (umol/L)
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 240 | 249
Micromoles per liter (umol/L) | 7.63 [6.46 to 8.80] | 1.12 [-0.03 to 2.27]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.51, 95% CI 2-sided [4.86 to 8.16]

12. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) From Creatinine Adjusted Using CKD-EPI Equation at Week 24
Description: Renal markers included GFR from creatinine adjusted using chronic kidney disease epidemiology collaboration (CKD-EPI) equation and summarized based on an OC data set at Week 24. Adjusted mean is the estimated mean change from Baseline in each biomarker at Week 24 in each arm calculated from an ANCOVA analysis of covariance model including the following covariates: treatment, original ART third agent class, interaction of treatment and original ART third agent class, and Baseline biomarker level. Differences are calculated as ABC/DTG/3TC - Current ART regimen.
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/second
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 240 | 249
mL/second | -8.05 [-9.30 to -6.80] | -1.18 [-2.41 to 0.06]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -6.87, 95% CI 2-sided [-8.64 to -5.11]

13. Secondary Outcome: Change From Baseline in GFR From Creatinine Adjusted Using MDRD Enzymatic Equation at Week 24
Description: Renal markers included GFR from creatinine adjusted using modification of diet in renal disease (MDRD) enzymatic equation and summarized based on an OC data set at Week 24. Adjusted mean is the estimated mean change from Baseline in each biomarker at Week 24 in each arm calculated from an ANCOVA analysis of covariance model including the following covariates: treatment, original ART third agent class, interaction of treatment and original ART third agent class, and Baseline biomarker level. Differences are calculated as ABC/DTG/3TC - Current ART regimen.
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/second/1.73 meter square
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 239 | 249
mL/second/1.73 meter square | -0.16 [-0.18 to -0.13] | -0.02 [-0.04 to 0.00]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.17 to -0.10]

14. Secondary Outcome: Change From Baseline in Urea at Week 24
Description: Renal markers included urea and summarized based on an OC data set at Week 24. Adjusted mean is the estimated mean change from Baseline in each biomarker at Week 24 in each arm calculated from an ANCOVA analysis of covariance model including the following covariates: treatment, original ART third agent class, interaction of treatment and original ART third agent class, and Baseline biomarker level. Differences are calculated as ABC/DTG/3TC - Current ART regimen.
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimoles per liter (mmol/L)
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 240 | 249
Millimoles per liter (mmol/L) | -0.03 [-0.18 to 0.12] | 0.07 [-0.08 to 0.22]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.375, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.31 to 0.12]

15. Secondary Outcome: Change From Baseline in Urine Albumin/Creatinine Ratio at Week 24
Description: Renal markers included urine albumin/creatinine ratioand summarized based on an OC data set at Week 24. Adjusted mean is the estimated mean change from Baseline in each biomarker at Week 24 in each arm calculated from an ANCOVA analysis of covariance model including the following covariates: treatment, original ART third agent class, interaction of treatment and original ART third agent class, and Baseline biomarker level. Differences are calculated as ABC/DTG/3TC - Current ART regimen.
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Gram per mole (G/mol) creatinine
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 197 | 222
Gram per mole (G/mol) creatinine | 0.11 [-0.70 to 0.92] | -0.07 [-0.84 to 0.69]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.749, ANCOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.93 to 1.30]

16. Secondary Outcome: Percent Change From Baseline in Bone Marker Analytes at Week 24
Description: Outcome Measure Description: Bone biomarkers analytes include bone specific alkaline phosphatase, osteocalcin, procollagen 1 n-terminal propeptide, type I collagen c-telopeptides and were analyzed based on log transformed data. Estimates were from an ANCOVA model adjusting for ART third agent class, interaction of treatment and original ART third agent class, age, sex (male or female), body mass index (BMI) (<25 kilogram per meter [kg/m] or >=25 kg/m), smoking status (never smoked or former smoker or current smoker), Baseline vitamin D (no vitamin D use at Baseline or vitamin D use at Baseline), and Baseline biomarker level.
Time Frame: Baseline and Week 24
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Percent
  Bone specific alkaline phosphatase, n= 214, 224 | 0.84 [0.79 to 0.88] | 0.98 [0.93 to 1.03]
  Osteocalcin, n=211, 221 | 0.87 [0.82 to 0.93] | 0.96 [0.90 to 1.03]
  Procollagen 1 n-terminal propeptide, n=212, 222 | 0.88 [0.83 to 0.94] | 0.96 [0.91 to 1.03]
  Type I collagen c-telopeptides, n=212, 223 | 0.87 [0.79 to 0.95] | 1.03 [0.94 to 1.14]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA — Bone specific alkaline phosphatase; Geometric Mean Ratio = 0.86, 95% CI 2-sided [0.82 to 0.90]
Statistical Analysis 2: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.002, ANCOVA — Osteocalcin; Geometric Mean Ratio = 0.91, 95% CI 2-sided [0.85 to 0.96]
Statistical Analysis 3: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.001, ANCOVA — Procollagen 1 n-terminal propeptide; Geometric Mean Ratio = -0.09, 95% CI 2-sided [-0.15 to -0.04]
Statistical Analysis 4: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.001, ANCOVA — Type I collagen c-telopeptides; Geometric Mean Ratio = 0.91, 95% CI 2-sided [0.86 to 0.96]

17. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analytes at Week 24
Description: Cardiovascular biomarkers were analyzed based on log transformed data. Estimates were from an ANCOVA model adjusting for ART third agent class, interaction of treatment and original ART third agent class, sex, race (white, black or African American, Other), and Baseline biomarker level.
Time Frame: Baseline and Week 24
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 276 | 277
Percent
  Fatty acid binding protein 2 [ng/L], n=212,222 | 0.67 [0.59 to 0.75] | 1.04 [0.92 to 1.17]
  Interleukin 6 [ng/L], n=213,222 | 0.86 [0.74 to 0.99] | 0.80 [0.69 to 0.92]
  Soluble cd14 [ng/L], n=214,223 | 0.76 [0.73 to 0.79] | 0.82 [0.79 to 0.85]
  Soluble vasc cell adhesion mol 1[ng/L], n=213,222 | 0.86 [0.80 to 0.92] | 0.85 [0.80 to 0.91]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA — Fatty acid binding protein 2; Geometric Mean ratio = 0.64, 95% CI 2-sided [0.57 to 0.72]
Statistical Analysis 2: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.311, ANCOVA — Interleukin 6; Geometric Mean ratio = 1.08, 95% CI 2-sided [0.93 to 1.24]
Statistical Analysis 3: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p < 0.001, ANCOVA — Soluble CD14; Geometric Mean ratio = 0.92, 95% CI 2-sided [0.89 to 0.96]
Statistical Analysis 4: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.742, ANCOVA — Soluble vasc cell adhesion molecule 1; Geometric Mean ratio = 1.01, 95% CI 2-sided [0.95 to 1.08]

18. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analyte, C-reactive Protein at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 226 | 231
Percent | 1.25 [1.04 to 1.50] | 1.25 [1.04 to 1.49]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.999, ANCOVA; Geometric Mean Ratio = 1.00, 95% CI 2-sided [0.84 to 1.19]

19. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analyte, D-Dimer at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 212 | 221
Percent | 1.00 [0.91 to 1.10] | 1.00 [0.91 to 1.10]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.981, ANCOVA; Geometric Mean Ratio = 1.00, 95% CI 2-sided [0.91 to 1.10]

20. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analyte, Homostat Model Assess of Insulin Resistance at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 210 | 219
Percent | 0.97 [0.84 to 1.11] | 1.00 [0.87 to 1.14]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.640, ANCOVA; Geometric Mean Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11]

21. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analyte, Insulin at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 213 | 222
Percent | 0.97 [0.86 to 1.09] | 0.99 [0.88 to 1.12]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.645, ANCOVA; Geometric Mean Ratio = 0.97, 95% CI 2-sided [0.87 to 1.09]

22. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analyte, Soluble CD163 at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 213 | 222
Percent | 1.09 [1.04 to 1.15] | 1.08 [1.02 to 1.13]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.577, ANCOVA; Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.97 to 1.06]

23. Secondary Outcome: Percent Change From Baseline in Cardiovascular Marker Analyte, Glucose at Week 24
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population. Only participants with a non-missing value at Week 24 are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 240 | 249
Percent | 1.02 [0.99 to 1.05] | 1.01 [0.99 to 1.04]
Statistical Analysis 1: Comparison: ABC 600 mg / DTG 50 mg /3TC 300 mg FDC vs Current ART; Test type: Superiority or Other; p = 0.687, ANCOVA; Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.98 to 1.03]

24. Secondary Outcome: Number of Participants With Incidence of Genotypic and Phenotypic Resistance Meeting Confirmed Virologic Withdrawal Criteria Over 24 Weeks
Description: Genotypic and phenotypic testing was conducted for participants who met the confirmed virologic withdrawal criteria, i.e., confirmed HIV-1 RNA >=400 c/mL any time after Day 1. The sample from the "suspected virologic withdrawal criterion" visit was tested for HIV-1 PRO and RT genotype and phenotype and HIV-1 integrase genotype and phenotype (i.e., the first of the two consecutive results >=400 c/mL). At the time of the data cut-off for this Week 24 analysis, no participants met the confirmed virologic withdrawal criteria over 24 weeks; therefore, the virologic analyses were not assessed.
Time Frame: Baseline and up to 24 weeks
Population: Viral Genotypic and Phenotypic Populations: Comprised of all participants in the ITT-E Population with available on-treatment genotypic and phenotypic resistance data, respectively, at the time confirmed virologic withdrawal criterion was met.
Arm/Group | ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Current ART
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Early Switch group AEs/SAEs are included from time of switch to ABC 600mg/DTG 50mg/3TC 300mg at baseline up to Week 48. Late Switch group AEs/SAEs are included from the time of switch to ABC 600mg/DTG 50mg/3TC 300mg at week 24 up to Week 48.
Description: Adverse events (AEs) and serious adverse events (SAEs) are presented for the early Switch and Late Switch group. AEs and SAEs were collected from participants of the safety population, comprised of all participants who received atleast one dose of the study drug.
Arm/Group | Early Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC | Late Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC
Serious Adverse Events (participants affected / at risk) | 9/275 | 6/244
Other Adverse Events (participants affected / at risk) | 101/275 | 61/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC (N=275) | Late Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC (N=244)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Homicide (Social circumstances) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Early Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC (N=275) | Late Switch ABC 600 mg / DTG 50 mg /3TC 300 mg FDC (N=244)
Diarrhoea (Gastrointestinal disorders) | 20 | 9
Upper respiratory tract infection (Infections and infestations) | 35 | 22
Nausea (Gastrointestinal disorders) | 28 | 15
Fatigue (General disorders) | 22 | 6
Headache (Nervous system disorders) | 17 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 6
Insomnia (Psychiatric disorders) | 14 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.